CLINICAL TRIAL: NCT05874349
Title: Histopathologic and Lymphocyte Subpopulations Evaluation of the Upper Gastrointestinal Tract of Crohn's Disease: A Multicentre Prospective Study (CROHNLY Project)
Brief Title: Histopathologic and Lymphocyte Subpopulations Evaluation of the Upper Gastrointestinal Tract of Crohn's Disease
Acronym: CROHNLY
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: CROHNLY23
Record Dates: First submitted 2023-04-12; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Crohn Disease
Keywords: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Crohn's disease: Patients with CD diagnosed according to the criteria of the ECCO guidelines. For the histological and lymphocyte subpopulation analysis of duodenal samples, all patients with CD who required an endoscopic examination during the disease have been prospectively included. All the recorded variables were registered at the moment of the endoscopy.
  Interventions: Behavioral: General variables; Behavioral: Clinical activity; Procedure: Laboratory data; Procedure: Endoscopic and histology data
- Cohort 2: Control groups: Two groups are included: 1) Disease control: Patients with celiac disease diagnosed according to the Catassi and Fasano criteria and 2) Healthy control subjects. For the histological and lymphocyte subpopulation analysis of duodenal samples, patients with celiac disease were prospectively included to undergone gastroscopy, before starting gluten-free diet. Control subjects were patients referred for upper endoscopy due to digestive symptoms that have normal appearing mucosa both at endoscopic and histological assessment (Marsh 0, <25 intraepithelial lymphocytes). Serological markers of celiac disease were negative and they have no signs of inflammatory bowel diseases.
  Interventions: Behavioral: General variables; Behavioral: Clinical activity; Procedure: Laboratory data; Procedure: Endoscopic and histology data

INTERVENTIONS:
Behavioral: General variables — Variables evaluated: age, sex, location, extent, and phenotype of IBD according to the Montreal classification, smoking habit, therapeutic requirements (immunosuppressants, biologics, steroids, salicylates, drugs that cause enteropathy such as olmesartan, valsartan, non-steroidal anti-inflammatory drugs, etc, ...).
Behavioral: Clinical activity — Clinical activity was evaluated using the Harvey-Bradshaw index (HBI) (cut-off values: <5, remission; 5-7, mild activity; 8-16, moderate activity; and >16, severe activity).
Procedure: Laboratory data — Laboratory data: blood count, renal function and C-reactive protein, anti-transglutaminase antibodies, genetic study of celiac disease DQ2.5, DQ8, and DQ2.2, study of parasites, fecal calprotectin.
Procedure: Endoscopic and histology data — Endoscopic signs suggestive of CD in UDT (presence of canker sores, ulcers, ...) and colon inflammatory activity was evaluated when available in patients with active disease using the Simple Endoscopic Score for CD (SES-CD: 0-2, remission; 3-6, mild endoscopic activity; 7-15, moderate endoscopic activity; and >15, severe endoscopic activity).
  Duodenal biopsies were assessed by 2 pathologists and were evaluated according to Marsh classification modified by Ensari [Marsh 0, 1, 2 or 3], the limit of normality for intraepithelial lymphocytes (IELs) per 100 enterocytes is set at 25, gastric biopsies (determination of H. Pylori by immunohistochemistry) and esophageal biopsies was recorded too.
  Percentage of lymphocyte subpopulations are assessed by flow cytometry.

SUMMARY:
Inflammatory bowel disease (IBD) comprises a series of disorders of unknown cause, such as ulcerative colitis (UC), Crohn's disease (CD) and indeterminate colitis (IC), associated with an over-the-top immune response that produces lesions of variable depth and extent in the intestine. They have a chronic course, without cure and with an unpredictable evolution. Clinical symptoms of CD are characterized by malaise, weight loss, fever, diarrhoea, abdominal pain, vomiting, sometimes palpable mass, perianal disease, among others. The disease is most frequently located in the ileocecal area, but all the entire digestive tract from the oral cavity to the rectum may be affected. The involvement of the upper gastrointestinal tract (UGT) (L4) in CD is frequently undiagnosed. From 1-7% of patients with CD refer symptoms or signs that are due to UG involvement. Chronic iron deficient anaemia, in the absence of digestive symptoms, is the only guiding sign that may alert about the diagnosis.

Furthermore, retrospective cohort studies suggest that CD of the UGT is associated with a worse prognosis. The systematic study of the UGT in the initial evaluation of CD at the time of diagnosis is not generally recommended in adulthood, European Crohn's and Colitis Organisation (ECCO) guidelines recommend upper endoscopy only if there are upper digestive symptoms (vomiting, dyspepsia, etc.). In the case of gastroscopy, gastric biopsies have to be performed due to the possible presence of focal active gastritis, which is considered very specific of CD. This statement is based on a limited series of cases published in 1980. On the other hand, systematic performance of duodenal biopsies is not recommended. This fact has caused that the histopathology of duodenal CD is very unknown and the need to perform duodenal biopsies of the UGT is still a matter of debate.

Macro and microscopic findings from the UGT have generally been used to differentiate between UC and CD in cases of IC. Among the macroscopic findings highlight the presence of sores or ulcers and most specific and frequent microscopic findings are granulomas and chronic inflammatory infiltrate respectively. However, it is known that CD can cause lymphocytic infiltration of the duodenal epithelium (duodenal lymphocytosis or lymphocytic enteritis) and villus atrophy. These are findings are characteristically found in celiac disease, and therefore, these histological lesions of the duodenum also propose the differential diagnosis between celiac disease and CD.

In addition, it must be considered that many of the patients with IBD take immunosuppressive for disease control, which have been reported to be the cause of lymphocytic enteritis and duodenal villus atrophy. This proposed drug-induced enteropathy is based only in a few series of cases in the context of treatment with azathioprine and methotrexate. There are no studies systematically evaluate how often these drugs can cause a "sprue like" enteropathy.

The lymphocytic enteritis of celiac disease has been associated with a specific pattern of lymphocyte subpopulations (increase in the percentage of CD3+TCRγẟ+ lymphocytes and decrease in the percentage of CD3-). It is unknown if CD duodenal lymphocytes is associated with a specific CD cytometric pattern. If so, the evaluation of lymphocyte subpopulations could be of great diagnostic aid when considering the differential diagnosis between celiac disease, CD and other forms of duodenal lymphocytosis.

DETAILED DESCRIPTION:
Hypothesis:

Routine evaluation of the upper digestive tract mucosa can be useful for the differential diagnosis between of adult CD and celiac disease, particularly in patients with chronic iron-deficient anemia and lymphocytic enteritis in the duodenum. The study of the lymphocytic subpopulations can help in the differential diagnosis of lymphocytic enteritis and identify in which cases are due to CD. Nowadays, the prevalence of "sprue-like" enteropathy associated with the use of immunosuppressants in CD is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Diagnosis of Crohn disease
* Diagnosis of Coeliac disease
* Control subjects
* Study period: The study period has been 36 months (June 2017 - June 2020)

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Pregnancy
* Serious comorbidities: heart disease, chronic obstructive pulmonary disease, liver disease, bleeding disorders, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The definition of the study population was patients with CD diagnosed according to the criteria of the ECCO guidelines. The definition of control populations was patients with celiac disease diagnosed according to the Catassi and Fasano criteria and control subjects.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Description of microscopic lesions in the upper digestive tract in patients with CD. | 3 years
  Microscopic duodenum lesions are measured by "Marsh classification modified by Ensari" of histologic findings:
  * Type 0: normal (<25 intraepithelial lymphocytes per 100 enterocytes).
  * Type 1: increased intraepithelial lymphocytes but no villous atrophy (>25 intraepithelial lymphocytes per 100 enterocytes).
  * Type 2: villi still present but shortened.
  * Type 3: complete villous atrophy.

SECONDARY OUTCOMES:
Percentage of lymphocyte subpopulations in the duodenum of patients with CD. | 3 years
  Percentage of lymphocyte subpopulations are assessed by flow cytometry.
Description of "sprue-like" enteropathy associated with the use of immunosuppressants in CD. | 3 years
  "sprue-like" enteropathy lesions are measured by "Marsh classification modified by Ensari" of histologic findings:
  * Type 0: normal (<25 intraepithelial lymphocytes per 100 enterocytes).
  * Type 1: increased intraepithelial lymphocytes but no villous atrophy (>25 intraepithelial lymphocytes per 100 enterocytes).
  * Type 2: villi still present but shortened.
  * Type 3: complete villous atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Esteve, PhD, MD, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No